CLINICAL TRIAL: NCT01946659
Title: Promoting Adherence to Sleep Apnea Treatment Through Health Education Among Blacks With Metabolic Syndrome
Brief Title: Promoting Adherence to Sleep Apnea Treatment Among Blacks With Metabolic Syndrome
Acronym: MetSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 09-193
Record Dates: First submitted 2013-02-05; First posted 2013-09-19 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Tailored Telephone Intervention
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adherence to Sleep Apnea Treatment (Experimental): The intervention arm of the study receives tailored education regarding Sleep Apnea by the study health educator via telephone.
  Interventions: Behavioral: Adherence to Sleep Apnea Treatment
- Standard Care Group (Other): The standard care group gets the standard print communications about sleep apnea produced by NLHBI and American Academy of Sleep Medicine.
  Interventions: Other: Standard Care Group

INTERVENTIONS:
Behavioral: Adherence to Sleep Apnea Treatment — A health education material prepared after focus group discussion with community leaders and patients would be administered to the participants with an experienced health educator through phone. Upto 10 calls per each patient will be made to either group until 6 months or the patient has a sleep test done.
  Other Names: Linguistically and culturally tailored intervention
  Arms: Adherence to Sleep Apnea Treatment
Other: Standard Care Group — The standard care group gets a standard print communications about sleep apnea produced by NLHBI and American Academy of Sleep Medicine
  Arms: Standard Care Group

SUMMARY:
This is a randomized controlled Trial to evaluate effect of a culturally and linguistically tailored, telephone-delivered behavioral intervention on adherence to recommended assessment and treatment of sleep apnea in Blacks with Metabolic Syndrome. The investigators believe low awareness of Sleep Apnea and the risk it imposes to an individual health plays an important role in underdiagnosis and low adherence to treatment among Blacks. Hence, culturally and linguistically tailored health education will decrease the knowledge gap and improve adherence to recommended assessment and treatment of sleep Apnea. the investigators believe the effect of adherence to treatment of Sleep apnea is shown to improve the components of Metabolic syndrome and hence promote well control of Hypertension, Diabetes, weight, triglyceride and cholesterol.

DETAILED DESCRIPTION:
Primary aim: To evaluate effect of a culturally and linguistically tailored, telephone-delivered behavioral intervention, versus an attention-control condition, on adherence to recommended assessment and treatment of sleep apnea.

Secondary aims: 1) To evaluate the maintenance of intervention effects on adherence 6 months post-intervention; and 2) To assess treatment effects on components of the metabolic syndrome (waist circumference, blood pressure, lipid level, and fasting plasma glucose/HbA1C).

Exploratory aim: To identify the mediators of adherence to recommended sleep apnea assessment and treatment following exposure to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* African American / carribean American / African.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Involvement with other study
* Unable to understand and sign the informed consent form
* Heart attack or stroke within the past 12 weeks
* Diagnosed with Obstructive Sleep Apnea and/or on treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change the knowledge of risk factors for sleep apnea and improve adherence to recommended assessment and treatment for sleep apnea. | 6 months
  The knowledge of risk factors for sleep apnea will be measured by the Apnea knowledge/Apnea beliefs Scale. The adherence to recommended assessment and treatment for sleep apnea will be measured by Continuos Positive Airway Pressure machine.

SECONDARY OUTCOMES:
Change in the components of metabolic syndrome (as measured by Hba1c, triglycerides, and Blood pressure) for those who adhered to the treatment of Sleep Apnea | 6 months
  Components of Metabolic syndrome include Hypertension, Diabetes, weight, triglyceride and cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean-Louis, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University, New York, New York, United States

REFERENCES:
- [Derived] Jean-Louis G, Newsome V, Williams NJ, Zizi F, Ravenell J, Ogedegbe G. Tailored Behavioral Intervention Among Blacks With Metabolic Syndrome and Sleep Apnea: Results of the MetSO Trial. Sleep. 2017 Jan 1;40(1):zsw008. doi: 10.1093/sleep/zsw008. PMID 28364475
- [Derived] Ramos AR, Wallace DM, Pandi-Perumal SR, Williams NJ, Castor C, Sevick MA, Mcfarlane SI, Jean-Louis G. Associations between sleep disturbances and diabetes mellitus among blacks with metabolic syndrome: Results from the Metabolic Syndrome Outcome Study (MetSO). Ann Med. 2015 May;47(3):233-7. doi: 10.3109/07853890.2015.1015601. Epub 2015 Apr 9. PMID 25856540
- [Derived] Williams NJ, Jean-Louis G, Brown CD, McFarlane SI, Boutin-Foster C, Ogedegbe G. Telephone-delivered behavioral intervention among blacks with sleep apnea and metabolic syndrome: study protocol for a randomized controlled trial. Trials. 2014 Jun 12;15:225. doi: 10.1186/1745-6215-15-225. PMID 24925227